CLINICAL TRIAL: NCT00320762
Title: Study of the Safety and Effectiveness of the Ologen (OculusGen) Collagen Matrix Implant as an Aid in Glaucoma and Pterygium Surgery
Brief Title: Ologen (OculusGen)-Glaucoma and Pterygium Historical Control Study in China Beijing Hospital
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pro Top & Mediking Company Limited (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mediking0501-2
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Glaucoma; Pterygium
Keywords: Glaucoma; Pterygium; collagen matrix; OculusGen; trabeculectomy; Anti scarring; pterygium recurrence; tissue engineering; Aeon Astron
MeSH Terms: conditions — Glaucoma; Pterygium

INTERVENTIONS:
Device: OculusGen Biodegradable Collagen Matrix Implant

SUMMARY:
The purpose of this study is to determine whether the OculusGen Collagen Matrix is effective and safe to implant as an aid of glaucoma and pterygium surgeries.

DETAILED DESCRIPTION:
ologen (OculusGen) Collagen Matrix is a porous, scaffold matrix. It is to be implanted on the top of the scleral flap and beneath the conjunctiva and Tenon's capsule at the end of trabeculectomy. The pores in the scaffold matrix range from 20 to 200µm, a size that is suitable for fibroblasts to grow randomly, through the body of the matrix without causing scarring. The space occupied by the collagen matrix scaffold creates room for the development of a filtration bleb. Immediately after implantation, the collagen matrix is absorbed with the aqueous humor that brings a certain pressure press on the top of the scleral flap which makes the dynamic balance for the aqueous system keep the IOP in the right side. The collagen matrix is bio-degraded within 90 days and will leave a physiologic space for the filtration bleb to facilitate control of intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Patient able to cooperate with study procedures and able to perform tests reliably
* Patient willing to sign informed consent
* Patient able and willing to complete postoperative follow-up requirements
* Glaucoma: one/both eye(s) is/are affected by glaucoma
* Pterygium: patient with pterygium

Exclusion Criteria:

* Known allergic reactions to collagen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
the effectiveness via the reduction of IOP and the incidence of pterygium recurrence | 180 day

SECONDARY OUTCOMES:
the safety via the incidence of complications and adverse events. | 180 day

CONTACTS AND LOCATIONS:
Overall Officials: Hong Dai, MD, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, China

REFERENCES:
- [Result] Hsu WC, Spilker MH, Yannas IV, Rubin PA. Inhibition of conjunctival scarring and contraction by a porous collagen-glycosaminoglycan implant. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2404-11. PMID 10937547